CLINICAL TRIAL: NCT05822089
Title: Comparison of Visual Outcomes of Enhanced Monofocal Intraocular Lenses
Brief Title: Intraindividual Comparison of EMO IOLs
Acronym: EMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Leydolt, Assoc. Prof. PD Dr, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1631/2021
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Age Related Cataracts
MeSH Terms: interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison of 7 groups receiving predefined monofocal and enhanced monofocal intraocular lenses (EMO IOLs). Investigated IOLs will be implanted subsequently according to the study protocol with one IOL type in the dominant eye and the other IOL type in the non- dominant eye.
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be masked to the intraocular lens implanted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Monofocal IOL I vs. enhanced monofocal IOL I (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm one (I) participants will receive a monofocal IOL (ZCB00) vs. an enhanced monofocal IOL (ICB00)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Monofocal IOL II vs. enhanced monofocal IOL I (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm two (II) participants will receive a monofocal IOL (Sensar 1AAB00) vs. an enhanced monofocal IOL (ICB00)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Monofocal IOL III vs. enhanced monofocal IOL II (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm three (III) participants will receive a monofocal IOL (Vivinex XY1)vs. an enhanced monofocal IOL (Vivinex Impress).
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Enhanced monofocal IOL II vs. enhanced monofocal IOL II (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm four (IV) participants will receive an enhanced monofocal IOL (Vivinex Impress) bilateral with a monovision target
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Monofocal IOL IV vs. enhanced monofocal IOL III (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm five (V) participants will receive an enhanced monofocal IOL (EnVista) vs. an enhanced monofocal IOL (LuxSmart)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Extended depth of focus IOL IV in eyes with low to moderate irregular astigmatism (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm six (VI) participants will receive an extended depth of focus IOL (Acrysof IQ Vivity) in both eyes if low to moderate irregular astigmatism is observed.
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Extended Depth of Focus IOL in eyes with irregular astigmatism (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm seven (VII) participants will receive an extended depth of focus IOL (IC-8 Apthera IOL) in one eye if irregular astigmatism is observed.
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Monofocal IOL IV vs. enhanced monofocal IOL IV (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm eight (VIII) participants will receive an enhanced monofocal IOL (EnVista) vs. an enhanced monofocal IOL (EnVista Aspire)
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Enhanced depth of focus IOL I vs. Enhanced depth of focus IOL I (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm nine (IX) participants will receive an enhanced depth of focus IOL (PureSee) bilateral with a monovision target.
  Interventions: Procedure: phacoemulsification and intraocular lens implantation
- Monofocal IOL VI and monofocal IOL III (Experimental): The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. In Arm ten (X) participants will receive a monofocal IOL (Vivinex XC1) bilateral or a monofocal IOL (Vivinex XY1) bilateral.
  Interventions: Procedure: phacoemulsification and intraocular lens implantation

INTERVENTIONS:
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (ZCB00) vs. an enhanced monofocal IOL (ICB00)
  Arms: Monofocal IOL I vs. enhanced monofocal IOL I
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (Sensar 1 AAB00) vs. an enhanced monofocal IOL (ICB00)
  Arms: Monofocal IOL II vs. enhanced monofocal IOL I
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (Vivinex XY1) vs. an enhanced monofocal IOL (Vivinex impress)
  Arms: Monofocal IOL III vs. enhanced monofocal IOL II
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of an enhanced monofocal IOL (Vivinex impress) in both eyes
  Arms: Enhanced monofocal IOL II vs. enhanced monofocal IOL II
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of an enhanced monofocal IOL (EnVista) vs. an enhanced monofocal IOL (LuxSmart)
  Arms: Monofocal IOL IV vs. enhanced monofocal IOL III
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of an extended depth of focus IOL (Acrysof IQ Vivity) in both eyes if low to moderate irregular astigmatism is observed
  Arms: Extended depth of focus IOL IV in eyes with low to moderate irregular astigmatism
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of an extended depth of focus IOL (IC-8 Apthera) in one eye if irregular astigmatism is observed
  Arms: Extended Depth of Focus IOL in eyes with irregular astigmatism
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (EnVista) vs. an enhanced monofocal IOL (EnVista Aspire)
  Arms: Monofocal IOL IV vs. enhanced monofocal IOL IV
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of an enhanced depth of focus IOL (PureSee) in both eyes
  Arms: Enhanced depth of focus IOL I vs. Enhanced depth of focus IOL I
Procedure: phacoemulsification and intraocular lens implantation — bilateral cataract surgery including phacoemulsification in individuals suffering from age-related cataract and intraocular lens implantation of a monofocal IOL (Vivinex XY1) in both eyes or a monofocal IOL (Vivinex XC1) in both eyes
  Arms: Monofocal IOL VI and monofocal IOL III

SUMMARY:
The investigational devices are approved intraocular lenses (IOLs) intended to be implanted after phacoemulsification in individuals suffering from age-related cataract with the need of cataract surgery. Cataract surgery with precedent bilateral randomized IOL implantation will be performed in subjects who have signed an informed consent form. Postoperative examinations will be implemented in accordance with the approved investigational plan.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract planned for phacoemulsification extraction and posterior IOL implantation
* Age 50 to 100
* Visual potential in both eyes of 20/25 or better as determined by investigators estimation
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Irregular Astigmatism (Acrysof IQ Vivity IOL, IC-8 Apthera IOL)
* postoperativ binocular best corrected distance visual acuity (BCVA) ≥ 1.0 decimal (Arm ten (X))
* Standard cataract surgery with bilateral implantation of a monofocal IOL (Vivinex XC1 or Vivinex XY1) (Arm ten (X))

Exclusion Criteria:

* Preceding intraocular surgery or ocular trauma
* Relevant other ophthalmic diseases that particularly effects the zonular apparatus (such as severe pseudoexfoliation syndrome, preceding cryocoagulation, trauma)
* Pupil diameter < 2.0 mm (photopic)
* Laser treatment
* Uncontrolled systemic or ocular disease
* Pregnancy/Nursing
* childbearing ability

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Distant corrected intermediate visual acuity | 2-6 months
  Primary outcome measure will be monocular distant corrected intermediate visual acuity (DCIVA) of each intraocular lens implanted. DCIVA will be assessed using standardized early treatment diabetic retinopathy study (EDTRS) charts on a logarithm of the minimum angle of resolution (logMAR) scale.
Best-corrected distance visual acuity (BCDVA) - Acrysof IQ Vivity IOL, IC-8 Apthera IOL | 3-5 months
  Primary outcome measure will be monocular best-corrected distance visual acuity (BCDVA) of each intraocular lens implanted in eyes with irregular astigmatism. BCDVA will be assessed using standardized early treatment diabetic retinopathy study (EDTRS) charts on a logarithm of the minimum angle of resolution (logMAR) scale.
Contrast sensitivity and reading ability - Vivinex XC1 and Vivinex XY1 | 2-6 months and 1-5 years
  Primary outcome measures for arm ten (X) will be the distance corrected contrast sensitivity and near corrected reading ability and reading speed. Contrast sensitivity will be assessed under standard photopic (85cd/m2) and mesopic (3cd/m2) conditions

SECONDARY OUTCOMES:
Contrast sensitivity and reading ability | 2-6 months and 1-5 years
  Secondary outcome measures will be the distance corrected contrast sensitivity and near corrected reading ability and reading speed. Contrast sensitivity will be assessed under standard photopic (85cd/m2) and mesopic (3cd/m2) conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Leydolt, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided